CLINICAL TRIAL: NCT06451952
Title: Virtual Darkness and Digital Phenotyping in Specialized and Municipal Dementia Care: The DARK.DEM Randomized Controlled Trial
Brief Title: Virtual Darkness Theraphy for Agitation in Dementia
Acronym: DARKDEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: NKS Olaviken Gerontopsychiatric Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFR sponsor code 334750; 697405 (Other: REK VEST (Ethical approval))
Record Dates: First submitted 2024-04-03; First posted 2024-06-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-11

CONDITIONS: Agitation in Dementia, Including Alzheimer's Disease
Keywords: virtual darkness theraphy; agitation in dementia; randomized controlled trial; gerontopsychiatric hospital
MeSH Terms: conditions — Aberrant Motor Behavior in Dementia

STUDY DESIGN:
Intervention Model Description: Open-label, single blinded randomized controlled trial, parallel arm, allocation ratio 1:1, to evaluate the superiority of virtual darkness as add on to treatment as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual darkness (Experimental): Exclusive exposure to light deprived of blue wavelengths from 19.00-08.00 for 14 consecutive days as add-on to treatment as usual (TAU). This will be provided in an ordinary part of the hospital ward with circadian lightening delivered by Chromawiso. This lightening is CE approved. The intervention will be delivered in two separate patient units, each of them will include one living room, one bedroom and a bathroom, area ranging from 58m2- 60 m2. If patients are able to wear blue blocking glasses (amber lenses), they can stay outside the units from 19.00-08.00. Between 08.00-19.00 the patients in the intervention groups can stay inside or outside the units as they wish.
  Interventions: Other: Virtual darkness
- Control condition (No Intervention): Treatment as usual for agitation in specialized dementia health services encompasses use of psychotropic drugs (anxiolytic agents, antipsychotic agents, antidementia agents), environmental interventions, music therapy and use of medical restraints

INTERVENTIONS:
Other: Virtual darkness — Chronotheraphy
  Arms: Virtual darkness

SUMMARY:
Behavioral and psychological symptoms of dementia (BPSD) such as anxiety, depression, psychosis and agitation, are prevalent, often treatment resistant, resource demanding and significantly deteriorates cognition, independency, quality of life and mortality in people with dementia.

The DARK.DEM trial aims at developing new diagnostics and treatment for BPSD in both specialized and municipal dementia care.

The investigators will develop digital phenotyping by determining the convergent validity of data from a smartwatch against established psychometric scales for BPSD for patients admitted to NKS Olaviken gerontopsychiatric hospital.

The investigators will conduct an open label single blinded randomized controlled trial to determine the effectiveness, feasibility and safety of virtual darkness as adjunctive treatment of agitation in patients with dementia admitted to the hospital. The investigators will randomize minimum 72 patients to treatment as usual (psychotropic drugs, psychological and environmental interventions) or 14 days of virtual darkness therapy, that is, exposure to light deprived of blue wavelengths from 19.00-08.00, provided in a secluded patient unit with circadian lightening. Primary outcome is 14 days change in agitation assessed with Cohen-Mansfield Agitation Inventory. Secondary outcomes are change in diurnal variation of motor activity assessed with a smartwatch and sleep monitor, other BPSD, activities of daily living, quality of life, use of psychotropic drugs, use of restraints and coercion, length of hospital stay and resource utilization.

The investigators will conduct focus group interviews with managers and staff in nursing homes to explore barriers, enablers and adaptions to support implementation of the new methods in municipal dementia care

DETAILED DESCRIPTION:
Successful treatment of BPSD relies on precise assessment. The gold standard is self-report of symptoms, supplemented by proxy rating from relatives and staff. This can be aided by various psychometric scales, such as the Cornell Scale for Depression, Cohen-Mansfield Agitation Inventory and Neuropsychiatric Inventory. However, these scales have weaknesses, they span short time periods, have moderate interrater and test-retest reliability. In particular in the outpatient setting, this hampers the reliability and validity of patients and caregivers reports, and thereby infers the accuracy of the clinicians assessment. A possible enhancement of assessment can be achieved through "digital phenotyping", that is characterization of human behavior by moment-by-moment monitoring with personal digital devices.

First line treatment of BPSD is environmental approaches, which often is resource demanding as it requires extensive staffing. Second line treatment is use of psychotropic drugs, however, effect is modest and come with high risk of interactions and side effects, particularly harmful in fragile older adults. A possible enhancement of BPSD treatment lies in interventions targeting the circadian rhythm. The circadian rhythm is weakened in persons with dementia, and this can potentiate BPSDs. Several trials have demonstrated some effect of bright light therapy on BPSD, however, it has been suggested that the effect is limited due to lack of sufficient light reaching the retina due to eye conditions in the elderly. Therefore, a more useful approach in this population might be virtual darkness, that is blue wavelength depleted evening light.

The DARK.DEM trials primary objective is to develop and evaluate digital phenotyping and virtual darkness therapy to enhance management of BPSD in municipal and specialized dementia care.

Secondary objectives are:

* Determine the feasibility of symptom assessment with wearable sensor technology in patients with dementia admitted to a gerontopsychiatric hospital ward.
* Determine the convergent validity of data obtained via sensor technology in patients with dementia against psychometric scales for assessment of BPSD.
* Determine the effectiveness, feasibility and safety of virtual darkness in the evening and night as adjunctive treatment of agitation in patients with dementia in a gerontopsychiatric hospital ward.
* Explore barriers, enablers and possible adaptions to support implementation of digital phenotyping and virtual darkness therapy in nursing homes.

The investigators will apply a multidisciplinary approach with methods from computer science, hermeneutics and medicine in three work packages (WP).

WP1: DIG.DEM will determine the convergent validity of sensor data against established psychometric scales for BPSD in patients admitted to NKS Olaviken gerontopsychiatric hospital. The investigators will use correlation analyses and knowledge based AI to develop novel digital biomarkers for BPSD.

WP2: DARK.DEM is an open label single blinded randomized controlled trial to determine the effectiveness, feasibility and safety of virtual darkness as adjunctive treatment of agitation in patients with dementia admitted to the hospital. The investigators will randomize minimum 72 patients to treatment as usual (psychotropic drugs, psychological and environmental interventions) or 14 days of virtual darkness therapy, that is, exposure to light deprived of blue wavelengths from 19.00-08.00, provided in a secluded patient unit with circadian lightening. Inclusion criteria is patients with dementia admitted to the hospital, both genders, above 50 years and CMAI score equal or above 45 points, exclusion criteria is total blindness/diminished bilateral red reflex, use of beta-blockers and/or melatonin, and clinically significant pain (MOBID-2 score equal or above 3 points). Primary outcome is 14 days change in agitation assessed with Cohen-Mansfield Agitation Inventory. Secondary outcomes are change in diurnal variation of motor activity assessed with sensor data, other BPSD, activities of daily living, quality of life, use of psychotropic drugs, use of restraints and coercion, length of hospital stay and resource utilization.

WP3: DECIDE.DEM will conduct focus group interviews with managers and staff in nursing homes to explore barriers, enablers and adaptions to support implementation of the new methods in municipal dementia care. The investigators will use a mixed methods explanatory sequential design, hermeneutical methodology.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to NKS Olaviken gerontopsychiatric hospital
* Diagnosis of dementia, all stages and etiologies,
* ≥50 years
* both genders
* Clinically significant agitation (CMAI ≥45)

Exclusion Criteria:

* Total blindness/diminished bilateral red reflex.
* Use of melatonin
* Clinically significant pain (MOBID-2≥3)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | Change from baseline to day 14
  The CMAI is a clinically validated agitation rating scale that measures the frequency of 29 items on agitated behaviors, encompassing four clusters of behavior: 1) aggressive behavior (e.g. hitting, kicking, screaming), 2) physically non-aggressive behavior (e.g. pacing, trying to get to a different place, restlessness), 3) verbally agitated behavior (complaining, constant requests for attention, repetitive questions) and 4) hiding and hoarding. Each of the 29 items are scored from 1 (no) to 7 (severe) evaluating the past 14 days. Scale range from 29-203, high score indicates severe symptoms. The CMAI correlates with other neuropsychiatric symptom scales, has high internal consistency and adequate inter-rater reliability with regard to physical aggression and verbal agitation.

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | Change from baseline to day 7
  The CMAI is a clinically validated agitation rating scale that measures the frequency of 29 items on agitated behaviors, encompassing four clusters of behavior: 1) aggressive behavior (e.g. hitting, kicking, screaming), 2) physically non-aggressive behavior (e.g. pacing, trying to get to a different place, restlessness), 3) verbally agitated behavior (complaining, constant requests for attention, repetitive questions) and 4) hiding and hoarding. Each of the 29 items are scored from 1 (no) to 7 (severe) evaluating the past 14 days. Scale range from 29-203, high score indicates severe symptoms. The CMAI correlates with other neuropsychiatric symptom scales, has high internal consistency and adequate inter-rater reliability with regard to physical aggression and verbal agitation.
Nevropsychiatric Inventory Nursing Home Version NPI-NH | Change from baseline to day 7, change from baseline to day 14
  Neuropsychiatric symptoms assessed with the Norwegian version of the Neuropsychiatric Inventory Nursing Home Version (NPI-NH): Instrument for proxy rating of neuropsychiatric symptoms in people with dementia over the past 4 weeks. A total of 12 items symptoms and behaviors are assessed regarding frequency (0: not present, 4: very frequent), severity (0: mild, 3: severe) and burden for caregivers (0: no burden, 5: severe burden), total score range 0-144, high score indicates frequent, severe and burdensome symptoms. The Norwegian version of NPH-NH has good validity and reliability
Cornell Scale for Depression in Dementia (CSDD) | Change from baseline to day 7, change from baseline to day 14
  Depressive symptoms assessed with Cornell Scale for Depression in Dementia (CSDD). This is an instrument for proxy rating of depressive symptoms in dementia over the past week. It has high inter-rater reliability, validity and sensitivity to change. A total of 19 symptoms are evaluated from 0= no symptoms to 2= severe symptoms. Total score range 0-38 points, score ≥8 indicates depression, score ≥ 12 indicates severe depression.
Sleep Disorder Inventory (SDI) | Change from baseline to day 7, change from baseline to day 14
  This instrument is an extended version of the one sleep item of the Neuropsychiatric Inventory (NPI) and proxy-rates sleep over the past 2 weeks. A total of 8 sleep behaviors are assessed regarding frequency (0: not present, 4: very frequent), severity (0: mild, 3: severe) and burden for caregivers (0: no burden, 5: severe burden), total score range 0-96, high score indicates frequent, severe and burdensome symptoms. In DARK.DEM, SDI will be used to evaluate sleep over the past 7 days
Confusion Assessment Method (CAM) | Change from baseline to day 7, change from baseline to day 14
  Delirium assessed with Confusion Assessment Method (CAM) short version. This instrument relies on staff observation to evaluate sudden start and fluctuation of symptoms, inattention, disorganized thoughts and awareness, each of these items are scored 1 if symptoms are present, high score indicated likely delirium. CAM has shown high sensitivity, specificity and inter-rater reliability in identifying delirium in samples with older adults and is also recommended for use in people with dementia.
Quality of life in dementia (QUALIDEM) | Change from baseline to day 7, change from baseline to day 14
  This instrument proxy rates the quality of life to persons with mild to severe dementia ≥65 years. The instrument structure and content are based on the adaption-coping model and covers nine domains of QoL: care relationship, positive affect, negative affect, restless tense behavior, positive self-image, social relations, social isolation, feeling at home and having something to do. A total of 40 items regarding behavior are evaluated according to frequency the last week (never, seldom, sometimes, often). The instrument has good reliability and validity.
Clinical Global Impression scale, CGI | Change from baseline to day 7, change from baseline to day 14
  Clinical impression A brief, stand-alone assessment of the clinician's view of the patient's global functioning prior and after an intervention and takes into account all available information, also including knowledge on the patient's history, psychosocial circumstances, symptoms, behavior and the impact of the symptoms on the patient's ability to function. CGI has two components 1) the Severity of illness (CGI-S): Considering the raters total clinical experience with this particular population, how mentally ill is the patient at this time rated on a seven-point scale from 1 (normal)-7 (most extremely ill patients). 2) Clinical Global Impression-Improvement (CGI-I) asks the clinician to compare the patients overall clinical condition to the one-week period to the initiation of the treatment: Compared to the patient's condition at baseline, this patient's condition is rated on a seven-point scale from 1 (very much improved) - 7 (very much worse)
Personal activities of daily living, P-ADL | Change from baseline to day 7, change from baseline to day 14
  This proxy rated instrument assess the ability to perform six areas of personal ADL, that is toileting, feeding, dressing, grooming, physical ambulation and showering, scale range 6-30, high score indicate worse outcome
Direct care time | Change from baseline to day 7, change from baseline to day 14
  Direct care time will be evaluated with assessment of how many hours/24 hours the staff provide care in 1 to 1 ratio, or 2 to 1 ratio (patient:staff ratio)
Use of drugs, numbers, use regularly | Change from baseline to day 7, change from baseline to day 14
  Drugs in use on day 7 and 14 will assessed from the participants medical journal and classified according to the ATC classification in numbers, use regularly
Use of drugs, doses, use regularly | Change from baseline to day 7, change from baseline to day 14
  Drugs in use on day 7 and 14 will assessed from the participants medical journal and classified according to the ATC classification in daily doses, use regularly
Use of drugs, numbers, use on demand | Change from baseline to day 7, change from baseline to day 14
  Drugs in use on day 7 and 14 will assessed from the participants medical journal and classified according to the ATC classification in numbers, use on demand
Use of drugs, doses, use on demand | Change from baseline to day 7, change from baseline to day 14
  Drugs in use on day 7 and 14 will assessed from the participants medical journal and classified according to the ATC classification in daily doses, use on demand
Decisions on coercion according the The Mental Health Act | Change from baseline to day 7, change from baseline to day 14, change baseline to until the date of discharge assessed up to 1 year
  Number of decisions
Decisions on coercion according the The Mental Health Act | Change from baseline to day 7, change from baseline to day 14, change from baseline to until the date of discharge assessed up to 1 year
  Type of decisions
Living situation | Change from baseline to until the date of discharge assessed up to 1 year
  Living situation at discharge categorized in at home- alone, at home- not alone, institution- temporary and institution- permanently
Length of hospital stay | Change from baseline to until the date of discharge assessed up to 1 year
  Length of hospital stay in days assessed from baseline to date of discharge.
Digital biomarker for agitation in dementia | Change from baseline to day 7, change from baseline to day 14
  Estimation of agitation in people with dementia resulting from digital measurements collected with the Empatica Embrace Plus wristband and Somnofy. Agitation is represented as a score defined over the interval 0-100, where 0 represents no agitation and 100 represents severe agitation (equivalent to maximum score on CMAI).
Digital biomarker for depression in dementia | Change from baseline to day 7, change from baseline to day 14
  Estimation of depression in people with dementia resulting from digital measurements collected with the Empatica Embrace Plus wristband and Somnofy. Depression is represented as a score defined over the interval 0-100, where 0 represents no depression and 100 represents severe depression (equivalent to maximum score on CSDD).
Digital biomarker for sleep in dementia | Change from baseline to day 7, change from baseline to day 14
  Estimation of sleep in people with dementia resulting from digital measurements collected with the Empatica Embrace Plus wristband and Somnofy. Sleep is represented as a score defined over the interval 0-100, where 0 represents no sleep disturbances and 100 represents severe sleep disturbances (equivalent to maximum score on SDI).
Digital biomarker for circadian rhythm in dementia | Change from baseline to day 7, change from baseline to day 14
  Estimation of circadian rhythm parameters in people with dementia resulting from digital measurements collected with the Empatica Embrace Plus wristband and Somnofy. The parameters are represented as a tuple of characteristics that together define the circadian rhythm.
Treatment emergent adverse events | Change from baseline to day 7, change from baseline to day 14
  Treatment Emergent Adverse Events will be evaluated in frequency and severity of headache, dizziness, depressive symptoms, eye strain, eye discomfort, blurred vision, falls, fractures, delirium, and the clinician evaluated causal relationship between the intervention and the serious adverse event (unlikely, possible, probable, definite). In addition, we will count the number of fractures, transference to somatic hospital and deaths

OTHER OUTCOMES:
Patient perspective (intervention group) | To be completed after day 14 of the intervention but before the date of discharge assessed up to 1 year
  Patient perspective: There is a lack in the literature on assessment tools to systematically evaluate a person with dementias perspective on treatment. Therefore, 3-5 questions will be developed to be evaluated by the person with dementia together with the responsible physician /psychologist after the intervention period (day 14). This could for example be: Have the participant noticed that it has received exposure to orange light during evening and night as supplemental treatment? (yes/no/partly) How did the participant perceive this light? (comfortable/uncomfortable/neutral/no opinion). How the participant perceive wearing a smartwatch? (invasive/not invasive/no opinion). This form will also have a blank space for quotations.

CONTACTS AND LOCATIONS:
Locations (1):
- NKS Olaviken Gerontopsychiatric Hospital, Askøy, Erdal, Norway

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: IPD will be shared with other researchers upon reasonable request to the principal investigator.